CLINICAL TRIAL: NCT00726505
Title: Characterization of the Kinetics of Renal Glucose Reabsorption in Response to Dapagliflozin in Healthy Subjects and in Subjects With Type 2 Diabetes Mellitus
Brief Title: Renal Mechanism of Action/Splay vs. TmG
Acronym: MOA
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MB102-020
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes, NOS
MeSH Terms: conditions — Diabetes Mellitus | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Active Comparator): Subjects with T2DM - Dapagliflozin 5 mg
  Interventions: Drug: Dapagliflozin
- Group 2 (Active Comparator): Subjects with T2DM - Dapagliflozin 20 mg
  Interventions: Drug: Dapagliflozin
- Group 3 (Active Comparator): Healthy Subjects - Dapagliflozin 20 mg
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Tablets, Oral, Once Daily, up to 29 days:
  Other Names: BMS-512148

SUMMARY:
The purpose of this study is to evaluate the effects of dapagliflozin to promote glucose loss in urine in healthy subjects and subjects with type 2 diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects
* Age 18 to 65 years
* BMI 18 to 35 kg/m2
* Healthy subjects and subjects with type 2 diabetes mellitus on 1 of the following therapies: diet, sulfonylurea, and/or metformin
* No evidence of impaired renal function

Exclusion Criteria:

* Unwilling or unable to use an acceptable method of birth control
* Subjects with type 1 diabetes mellitus, heart disease, hepatic C or B
* Exposure to insulin
* Use of exclusionary concomitant medications
* Evidence of significant kidney disease or any other significant medical or psychiatric disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The change in urinary glucose excretion dynamics | after 7 days of treatment

SECONDARY OUTCOMES:
Differences in urinary glucose between healthy and diabetic subjects | at 7 days
Changes in liver glucose production | at one day
Glucose effects on tubular markers | at one day

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- University Of Texas Health Center At San Antonio, San Antonio, Texas, United States

REFERENCES:
- See also: MB102020 _Redacted _CSR _synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3635&filename=MB102020%20_Redacted%20_CSR%20_synopsis.pdf